CLINICAL TRIAL: NCT07275840
Title: An Open-label, Multicenter, Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of Intravitreal Injection of IBI302 in Participants With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Evaluate the Efficacy and Safety of IBI302inSubjects With nAMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI302A203
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — IBI302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI302 8mg dose 8mg (Experimental): Drug: IBI302 8mg/Intravitreal injection
  Interventions: Drug: IBI302 8mg dose

INTERVENTIONS:
Drug: IBI302 8mg dose — 8 mg IBI302 will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by once every 8 weeks.

SUMMARY:
This study is designed for Open-label, multi-center, single-arm Phase II trail to evaluate the efficacy and safety of intravitreal injection of IBI302 in nAMD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an informed consent form before participating in the research.
2. Male or female individuals aged 50 or above at the time of signing the informed consent form;
3. Active CNV under the macular fovea secondary to nAMD or active CNV involving the macular fovea.
4. At baseline, the BCVA of the study eye was within the range of 19 to 78 ETDRS letters (including both ends).

Exclusion Criteria:

1. According to the investigator's judgment, concomitant ocular diseases/systemic diseases of the study eyes at screening or baseline may lead to participants' non-response to the study treatment or confuse the interpretation of the study results;
2. The study eye has uncontrollable glaucoma;
3. There is an active intraocular or periocular infection or inflammation in either eye;
4. The non-study eye has severe visual function disorders;
5. Within 90 days before baseline, the study eye had received anti-VEGF treatment;
6. Within 90 days before baseline, the study eye had received anti-complement treatment;
7. At any time before baseline, the study eye had received IBI302 treatment;
8. Uncontrollable hypertension;
9. Glycated hemoglobin (HbA1c) > 10.0% within 28 days prior to screening;
10. Other exclusion criteria set by protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants whose best corrected visual acuity (BCVA) of the study eye decreased by less than 15 letters from baseline as measured by the visual acuity chart in the early treatment diabetic retinopathy study (ETDRS) at week 52 | Week52

SECONDARY OUTCOMES:
The changes in BCVA from baseline at each visit | Baseline，Weeks 4，8，12，16，20，24，28，32，36，40，44，48 and 52
Proportion of patients with BCVA improvement of ≥0, ≥5, ≥10, and ≥15 ETDRS letters from baseline at week 52 | Week52
Proportion of participants with a decrease in BCVA of >0, ≥5, ≥10, and ≥15 ETDRS letters from baseline at week 52 | Week52
The change in central subfield thickness of the macula measured by OCT from the baseline at week 52 | Week52
Proportion of participants with IRF/SRF/Pigment epithelial detachment (PED) on OCT at Week 52 | Week52
Change in choroidal neovascularization (CNV) area on fundus fluorescein angiography (FFA) at week 52 compared to baseline | Week52
Change in CNV leakage area on FFA at week 52 compared to baseline | Week52
Proportion of participants with new-onset MA on OCT at Week 52 | Week52
Proportion of new-onset fibrosis on color fundus photography (CFP) at Week 52 | Week52
Change in MA area on OCT from baseline at Week 52 | Week52
Change in fibrosis area and maximum lesion diameter on CFP from baseline at Week 52 | Week52
The incidence rate, correlation with the studied drugs, and severity of ocular and systemic adverse events (AE), treatment emergent adverse events (TEAE), and serious adverse events (SAE) | From baseline through Week 52
The production of anti-drug antibodies in the serum | Day0、Week4、Week16、Week32、Week48、Week52

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai general hospital, Shanghai, Shanghai Municipality, China